CLINICAL TRIAL: NCT00742170
Title: Transdermal Electroacupuncture for Opioid Detoxification
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Scott Lukas, Pharmacologist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-P000711
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Opioid Dependency
Keywords: opioid dependence; opioid detoxification; electroacupuncture; adjunctive treatment; alternative/complementary medicine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active electroacupuncture (Active Comparator): In the active electroacupuncture condition, the current is set at 2 times threshold (approximately 6-10 mA), which typically produces muscle twitching.
  Interventions: Device: Electroacupuncture
- Sham electroacupuncture (Sham Comparator): In the sham electroacupuncture condition, the current is set at 1 mA, the lowest intensity possible before the HANS device shuts off; this is undetectable stimulation.
  Interventions: Device: Electroacupuncture

INTERVENTIONS:
Device: Electroacupuncture — Participants are randomly assigned to receive either active or sham electroacupuncture using the Han's Acupoint Nerve Stimulator (HANS) device. The HANS method uses a non-invasive device that emits a constant electric current transcutaneously via skin electrodes to stimulate relevant acupoints: Heku (LI4) / Laogong (P8) on one hand and Neiguan (P6) / Waiguan (TE 5) on the opposite arm. Stimulation is delivered in the dense-and-disperse mode, alternating between 2 and 100 Hz at 3-second intervals. Participants receive thrice daily treatments for 4 days during inpatient opioid detoxification.

SUMMARY:
This single-blind, randomized clinical trial tests whether electroacupuncture, provided as an adjunctive treatment, improves outcomes among patients receiving inpatient opioid detoxification from opioids.

DETAILED DESCRIPTION:
Opioid dependence continues to be a major public health concern in the United States, with prescription opioid abuse rapidly becoming one of the nation's biggest drug problems. Although there have been substantial improvements in the pharmacological treatment of opioid dependence, many patients relapse soon after detoxification. In China and other countries, acupuncture has been effective in the treatment of heroin dependence. The current study tests whether electroacupuncture, provided as an adjunctive treatment, produces improved outcomes among patients receiving inpatient detoxification from opioids. The primary hypothesis is that participants who receive active electroacupuncture, compared to those receiving sham electroacupuncture, will experience milder withdrawal symptoms, report less opioid craving, and maintain abstinence from opioids for longer duration following discharge. This study will be a single-blind, randomized clinical trial in which participants will receive either active or sham electroacupuncture. Participants will be recruited from the inpatient unit at the Alcohol and Drug Abuse Treatment Program at McLean Hospital. Participants will receive thrice daily 30-minute electroacupuncture treatments for 4 days. The Han's Acupoint Nerve Stimulator device will be used to stimulate acupoints on one hand (LI4/P8) and opposite arm (P6/TE5). This device emits a constant electric current transcutaneously via skin electrodes to stimulate relevant acupoints. It does not use needles and has no harmful side-effects. Participants will be followed for 2 weeks following discharge. Assessments will occur daily during the treatment phase and weekly during the follow-up phase. Assessments will include clinical interviews, questionnaires, urine toxicology screens, and medical record review. The results of this study will indicate whether short-term electroacupuncture may be of benefit to individuals receiving inpatient detoxification from opioids.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid dependence
* Current buprenorphine detoxification
* 18-59 years of age
* English proficiency

Exclusion Criteria:

* Acute mania, psychosis, or suicidality
* Cognitive impairments precluding informed consent
* Heart disease or contraindicated heart condition
* Use of pace maker
* History of seizure disorder
* Current detoxification from alcohol or benzodiazepines
* Inability to return to follow-up visits
* For women, pregnancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Lukas, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Meade CS, Lukas SE, McDonald LJ, Fitzmaurice GM, Eldridge JA, Merrill N, Weiss RD. A randomized trial of transcutaneous electric acupoint stimulation as adjunctive treatment for opioid detoxification. J Subst Abuse Treat. 2010 Jan;38(1):12-21. doi: 10.1016/j.jsat.2009.05.010. Epub 2009 Jul 1. PMID 19574017

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Electroacupuncture Condition: Active electroacupuncture condition
  Electroacupuncture: Participants are randomly assigned to receive either active or sham electroacupuncture using the Han's Acupoint Nerve Stimulator (HANS) device. The HANS method uses a non-invasive device that emits a constant electric current transcutaneously via skin electrodes to stimulate relevant acupoints: Heku (LI4) / Laogong (P8) on one hand and Neiguan (P6) / Waiguan (TE 5) on the opposite arm. Stimulation is delivered in the dense-and-disperse mode, alternating between 2 and 100 Hz at 3-second intervals. Participants receive thrice daily treatments for 4 days during inpatient opioid detoxification.
- Sham Electroacupuncture Condition: In the sham electroacupuncture condition, the current is set at 1 mA, the lowest intensity possible before the HANS device shuts off; this is undetectable stimulation.
  Electroacupuncture: Participants are randomly assigned to receive either active or sham electroacupuncture using the Han's Acupoint Nerve Stimulator (HANS) device. The HANS method uses a non-invasive device that emits a constant electric current transcutaneously via skin electrodes to stimulate relevant acupoints: Heku (LI4) / Laogong (P8) on one hand and Neiguan (P6) / Waiguan (TE 5) on the opposite arm. Stimulation is delivered in the dense-and-disperse mode, alternating between 2 and 100 Hz at 3-second intervals. Participants receive thrice daily treatments for 4 days during inpatient opioid detoxification.
Period: Overall Study
Arm/Group | Active Electroacupuncture Condition | Sham Electroacupuncture Condition
Started | 26 | 29
Completed | 24 | 24
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Active Stimulation: In the active electroacupuncture condition, the current is set at 2 times threshold (approximately 6-10 mA), which typically produces muscle twitching.
  Electroacupuncture: Participants are randomly assigned to receive either active or sham electroacupuncture using the Han's Acupoint Nerve Stimulator (HANS) device. The HANS method uses a non-invasive device that emits a constant electric current transcutaneously via skin electrodes to stimulate relevant acupoints: Heku (LI4) / Laogong (P8) on one hand and Neiguan (P6) / Waiguan (TE 5) on the opposite arm. Stimulation is delivered in the dense-and-disperse mode, alternating between 2 and 100 Hz at 3-second intervals. Participants receive thrice daily treatments for 4 days during inpatient opioid detoxification.
- Sham Stimulation: In the sham electroacupuncture condition, the current is set at 1 mA, the lowest intensity possible before the HANS device shuts off; this is undetectable stimulation.
  Electroacupuncture: Participants are randomly assigned to receive either active or sham electroacupuncture using the Han's Acupoint Nerve Stimulator (HANS) device. The HANS method uses a non-invasive device that emits a constant electric current transcutaneously via skin electrodes to stimulate relevant acupoints: Heku (LI4) / Laogong (P8) on one hand and Neiguan (P6) / Waiguan (TE 5) on the opposite arm. Stimulation is delivered in the dense-and-disperse mode, alternating between 2 and 100 Hz at 3-second intervals. Participants receive thrice daily treatments for 4 days during inpatient opioid detoxification.
- Total: Total of all reporting groups
Arm/Group | Active Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (8.9) | 27.0 (8.6) | 27.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 18 | 21 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 23 | 28 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Using Drugs
Time Frame: 2 weeks following discharge
Measure: Number; unit: percent
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 17 | 17
percent | 35 | 77

2. Secondary Outcome: Opioid Craving (Self-report)
Description: Self-report on scale of 3 to 30 (higher number indicates more craving)
Time Frame: at 2-weeks post discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 17 | 17
units on a scale | 10.7 (7.2) | 14.3 (6.9)

ADVERSE EVENTS:
Arm/Group | Active Stimulation | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 0/26 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No